CLINICAL TRIAL: NCT06986213
Title: Heart Pillow - Chemoteraphy
Acronym: Hepi_Qt
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: José Manuel Afonso Moreira (Other)
Collaborators: Unidade Local de Saúde do Alentejo Central (Unknown); University of Évora (Other)
Responsible Party: Sponsor-Investigator, José Manuel Afonso Moreira, Clinical Professor, University of Évora
Organization: University of Évora (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: University of Évora-ULSAC
Record Dates: First submitted 2025-04-16; First posted 2025-05-22 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Rehabilitation Program; Breast Cancer Patients
Keywords: Breast cancer; nursing rehabilitation care; self-care; upper limb
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Participants are assessed using the instruments and techniques already mentioned. The data are analyzed from a clinical perspective to define and validate diagnoses. Validation is carried out by a rehabilitation nursing specialist. The diagnoses are in accordance with the International Classification for Nursing Practice:
  - Committed eating self-care. Self-care transfer committed Self-care grooming (toilet) committed Compromised self-care (going to the bathroom, bladder and bowel control) Compromised hygiene self-care Self-care walking (mobility and going up/down stairs), compromised Inadequate scar tissue The intervention is teaching and training with assistive devices for self-care and teaching and training in massage technique.
  Progress monitoring is carried out every 2 or 3 weeks, coinciding with the chemotherapy treatment plan.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Heart Pillow Group (Experimental)
  Interventions: Behavioral: Heart Pillow Intervention

INTERVENTIONS:
Behavioral: Heart Pillow Intervention — Self-Care:
  Teach techniques to perform diminished or dependent self-care. Demonstrate assistive devices for self-care. Teach and train techniques and the use of assistive devices.
  Scare Tissue:
  Perform massage techniques on scar tissue: gliding and friction. Teach and train massage technique.

SUMMARY:
Breast cancer is a health problem with increasing prevalence, along with more effective therapeutic responses and less mutilating surgeries. The process of caring for patients crosses different levels: the diagnostic phase, which is mostly outpatient, the surgical treatment phase, which is mostly short-term inpatient, and the medical treatment phase in a day hospital. An integrated and structured care model based on specialized nursing skills can help improve self-care, quality of life and well-being.

DETAILED DESCRIPTION:
Detailed description 1:

The intervention project is developed during the medical treatment phase and is designed to reconcile multidisciplinary interventions and accompany patients during this phase. Self-care is the central concept of the project, it is multidimensional but the approach in the project is centered on a disease process and people-centered healthcare responses. It is estimated that the early initiation of activities that promote the recovery of self-care and the reduction of complications resulting from immobility of the homolateral upper limb or the formation of scar adhesions may reduce the time and costs dedicated to rehabilitation care at a later stage.

The study includes personalized interventions, carried out with patients every three weeks, from the beginning until discharge from chemotherapy treatment. Once informed consent has been obtained, the first session carried out by the rehabilitation nurse includes the patient's assessment, the allocation of the Heart pillow with a teaching session and training for its use. The first assessment includes: sociodemographic and health characterization, assessment of symptoms and quality of life (EORTC QLQ-C3 version 3.0 and EORTC QLQ-Br23), independence in ADL (Barthel Scale), upper limb functionality (DASH Portuguese version), sleep quality (PSQI-PT), assessment of grip strength by dynamometry (Dynamometry), assessment of the range of movement of the upper limbs by goniometry and assessment of the presence of edema by measuring the limb circumference. The data collected at this stage are analyzed from a clinical perspective to define the individual care plan: Intervention in self-care and the symptoms mentioned.

Every 3 weeks, the assessment of symptoms, independence of daily activities, strength, range of movement and lymphedema are repeated, providing data on progress but also for assessing the individual care plan from which teaching and training interventions are carried out, appropriate for each participant.

The final assessment coincides with the completion of the last chemotherapy treatment session, the assessments of the intermediate phase are repeated and independence in instrumental activities and sleep quality are assessed.

Objectives:

Analyze the effects of the Heart Pillow in relieving symptoms. Analyze the results of self-care teaching and training in the recovery of functional independence of breast cancer patients treated with surgery, during chemotherapy treatment.

Characterize the evolution of symptoms during chemotherapy treatment.

Detailed Description 2:

Patient participation is obtained through informed consent. The heart-shaped pillow is supplied with a user manual and instructions are provided on how to use it. The manual was created by researchers, based on the results of the impact study with 93 women (awaiting publication).

After surgery and the resumption of chemotherapy treatments, participants are evaluated in the office (privacy and confidentiality) with the application of scales and questionnaires validated for the population studied and with techniques by a specialist in rehabilitation nursing (Goniometry and dynamometry) and evaluation of the surgical scar.

The EORTC QLQ-C3 version 3.0 and EORTC QLQ-Br23 questionnaires assess the presence and intensity of symptoms associated with breast cancer treatment and also the perception of quality of life. The Barhtel index provides data on the patient's independence in 10 activities of daily living (self-care). The Portuguese version of DASH identifies activities that are limited in the upper limb ipsilateral to the surgery. Sleep quality (PSQI-PT) is a study variable that emerged from research findings on the impact of pillows on women's symptoms and well-being. Data on sleep quality are collected at the beginning and end of the study.

Muscle strength, range of motion in the upper limb, and scar status are physiological variables that may be altered and may underlie limitations or dependence in performing self-care.

Chemotherapy treatment is performed every 3 weeks and assessments are also repeated with: Barthel Index, EORTC QLQ-C3 version 3.0 and EORTC QLQ-Br23, DASH, dynamometry, goniometry and scar assessment.

In all assessments, nursing diagnoses are defined and validated in accordance with the International Classification for Nursing Practice. The assessment data is analyzed and validated by experts to attest to its adequacy. For each diagnosis, an intervention plan is created that includes demonstration of techniques and support devices for self-care with a moderate or severe degree of dependence, teaching and training in techniques and use of devices. In the presence of the diagnosis of "Inadequate scar tissue" the intervention plan includes demonstration, teaching and training of massage technique.

At the end of chemotherapy treatment, the entire initial assessment is repeated. The data is recorded on specific, coded forms, and the information is transferred to an encrypted computer file, with access restricted to researchers. The file is destroyed after the study data has been published and disseminated.

ELIGIBILITY:
Inclusion Criteria:

* Breast cancer patients undergoing chemotherapy after surgery.

Exclusion Criteria:

* Patients with breast cancer who did not undergo surgical treatment.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Recovering mobility in the homolateral upper limb | Every 3 weeks until the end of chemotherapy treatment. The result of the evaluation is translated into: Kgf (Muscle strength); Degrees (goniometry). Time Points: T0-first evaluation appointment (chemotherapy); T1 at Tx-evaluation every 3 weeks
  The measures used are functional assessment of the upper limb with the Disabilities of the Arm, Shoulder and Hand (DASH-PT) scale: 30-item self-reported questionnaire in which the response options are presented as 5-point Likert scales. Scores range from 0 (no disability) to 100 (most severe disability). Assessment of muscle strength with dynamometry and assessment of amplitude by goniometry.

OTHER OUTCOMES:
Upper limb lymphoedema | Every 3 weeks until the end of chemotherapy treatment. Time Points: T0-first evaluation appointment (chemotherapy); T1 at Tx-evaluation every 3 weeks
  The measures used are assessment by palpation and observation of scar tissue. The result of the lymphoedema assessment translated into: centimeters
Sleep quality | At the start of chemotherapy after surgery, until the end of the treatment cycle (approximately 3 months). Time Points: T0-first evaluation appointment (chemotherapy); T1 at Tx-evaluation every 3 weeks
  The measure used is the Pittsburgh Sleep Quality Index (PSQI-PT) questionnaire. The PSQI consists of 19 items (plus 5 clinically relevant questions not considered for scoring purposes), which are distributed into seven "components": subjective sleep quality; sleep latency; sleep duration; habitual sleep efficiency; sleep disturbances; use of sleeping medication; day-time dysfunction. Each component is scored from 0 a 2, and the sum of the component scores yields a global PSQI score.

CONTACTS AND LOCATIONS:
Overall Officials: Isabel Bico, PhD, Principal Investigator — University of Évora; Paula Sousa, MsC, Study Chair — ULSAC; Sofia Braga, MsC, Study Chair — ULSAC; Carmelinda Talhinhas, Study Chair — ULSAC; José Moreira, Study Chair — University of Évora
Locations (1):
- Évora, Evora, Portugal

IPD SHARING:
Plan to Share IPD: No
Participants' personal data will not be shared, as recommended by the ethics committee. All data will be anonymized.

REFERENCES:
- See also: Related Info — https://gco.iarc.fr/today/en/dataviz/maps-heatmap?mode=population
- See also: Related Info — https://doi.org/10.5772/intechopen.108946